CLINICAL TRIAL: NCT07193121
Title: Effects of Wrestling Training on Psychological Well-Being, Anxiety, and Resilience in Adolescent Boys
Brief Title: Effects of Wrestling Training on Psychological Well-Being, Anxiety, and Resilience in Adolescent Sedanter Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/06
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Performance Enhancement; Supportive Care
Keywords: combat sports; psychological resilience; well-being; anxiety; mental health
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Model Description The statistical framework of the study was based on a two-way repeated-measures analysis of variance (ANOVA) designed to evaluate the effects of the wrestling intervention over time while accounting for within-subject and between-group variability.
  Model Structure
  The analytic model included:
  Within-subject factor:
  Time (2 levels: Pre-test, Post-test)
  Between-subject factor:
  Group (2 levels: Wrestling Group, Control Group)
  This produced a 2 × 2 mixed-model design, allowing the evaluation of:
  Main effect of Time Indicates whether psychological variables changed across the entire sample from pre- to post-test.
  Main effect of Group Tests whether the groups differed overall, independent of time. Group × Time interaction The primary parameter of interest, indicating whether the pattern of change over time differed between groups.
  Model Assumptions
  The repeated-measures ANOVA relied on the following assumptions:
  Normality:Shapiro-Wilk test. Homogeneity of Variance; Spherici
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wrestling training Group (Experimental): Both groups underwent baseline assessments before the intervention and post-tests after six weeks. The Wrestling Group participated in a structured wrestling training program, while the Control Group maintained their usual daily routines without additional exercise.
  Interventions: Other: Wrestling Group; Device: Control
- CONTROL (No Intervention): Control

INTERVENTIONS:
Other: Wrestling Group — Both groups underwent baseline assessments before the intervention and post-tests after six weeks. The Wrestling Group participated in a structured wrestling training program, while the Control Group maintained their usual daily routines without additional exercise.
  Arms: wrestling training Group
Device: Control — No intervention
  Arms: wrestling training Group

SUMMARY:
This randomized controlled study investigated the psychological effects of a six-week, non-competitive wrestling training program in sedentary adolescent boys. Thirty participants were assigned to either a wrestling group or a control group. Psychological well-being (WHO-5), sport anxiety (SAS-2), and resilience (BPRS) were measured before and after the intervention.

The wrestling group showed significant improvements in well-being and psychological resilience, along with marked reductions in total sport anxiety and its subcomponents (worry, somatic anxiety, concentration disruption). All changes demonstrated large effect sizes, while the control group exhibited no meaningful positive changes.

Overall, the findings suggest that even short-term, structured wrestling training can enhance emotional well-being, reduce anxiety, and strengthen resilience in adolescent boys. The study highlights wrestling as a promising physical activity for supporting youth mental health.

DETAILED DESCRIPTION:
Detailed Description of the Study Purpose and Rationale The study explores how short-term wrestling training affects psychological well-being, anxiety, and resilience in adolescent boys. While the physical benefits of wrestling are well known, its psychological impacts-especially in non-competitive, beginner contexts-have been insufficiently studied. Adolescence is a critical developmental period marked by heightened emotional sensitivity and vulnerability to stress and anxiety. Given the known mental health benefits of structured physical activity, the authors aimed to determine whether wrestling could serve as a mental health-supportive intervention for youth.

Study Design and Participants

The research employed a randomized controlled pretest-posttest design involving 30 sedentary male adolescents aged 12-15 years. Participants were divided into:

Wrestling Group (n = 15) Control Group (n = 15) Inclusion criteria ensured no prior experience with wrestling or other combat sports and minimal physical activity in the preceding six months. The study was ethically approved and conducted following the Declaration of Helsinki.

Intervention The wrestling group completed a six-week structured wrestling program with sessions three times per week, each lasting 60 minutes. The program progressed through foundational stances, entries, defensive techniques, agility, strength drills, and integrated combined training sessions. Warm-ups, dynamic stretching, and wrestling-specific drills formed each session's core. All sessions were supervised by certified coaches, with 100% adherence and no injuries.

The control group maintained their daily routines without added exercise.

Measurements

Three validated psychological scales were used:

WHO-5 Well-Being Index Measures positive mood and general well-being.

Sport Anxiety Scale-2 (SAS-2)

Includes subscales for:

Worry Somatic Anxiety Concentration Disruption Brief Psychological Resilience Scale (BPRS) Evaluates ability to recover from stress. Assessments were conducted at baseline and post-intervention under standardized laboratory conditions.

Statistical Analysis Data normality was examined with the Shapiro-Wilk test. A two-way repeated-measures ANOVA evaluated group × time interactions, with Bonferroni post-hoc tests where necessary. Partial eta squared (ηp²) quantified effect sizes, interpreted based on established benchmarks.

Key Findings

1. Psychological Well-Being The wrestling group showed a significant increase in WHO-5 well-being scores. The control group showed no significant change. The effect size was large (ηp² = 0.717).
2. Sport Anxiety

   Overall sport anxiety and all its subcomponents exhibited significant changes:

   Worry Wrestling group: significant decrease Control group: significant increase Somatic Anxiety Significant decreases in both groups, though greater in the wrestling group. Concentration Disruption Wrestling group: significant decrease Control group: significant increase Total Sport Anxiety Wrestling group: strong reduction Control group: strong increase Effect size extremely large (ηp² = 0.938)
3. Psychological Resilience Wrestling group: significant improvement Control group: no change Effect size: ηp² = 0.519 Interpretation of Results

The data indicate that structured, non-competitive wrestling training:

Enhances emotional well-being Reduces both cognitive and physical symptoms of anxiety Supports the development of resilience and stress recovery abilities Helps maintain concentration and reduce performance-related worry These findings align with prior research showing psychological benefits of combat sports, such as improved self-control, emotional regulation, and coping strategies.

The simultaneous increase in anxiety in the control group suggests that adolescence alone may contribute to rising stress levels-highlighting the protective role of physical activity.

Practical Implications

The study provides evidence that wrestling, even at a beginner level, can serve as:

A preventive mental health intervention A structured environment that promotes emotional stability A method to build psychological resilience in adolescent boys A supportive physical activity option for school and community programs The influence appears beneficial even within six weeks, without competitive pressures.

Limitations Small sample size (n = 30) Only male adolescents Conducted within a single cultural context Short intervention duration No long-term follow-up Future studies should investigate long-term effects, gender differences, hormonal or neurophysiological mechanisms (e.g., cortisol, HRV), and comparisons with other sports.

Conclusion The study demonstrates that a six-week wrestling training program significantly improves psychological well-being and resilience while reducing sport-related anxiety in adolescent boys. These findings support the potential of wrestling as a valuable tool for promoting youth mental health in structured, safe, non-competitive environments.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescents aged 12-15 years
* Sedentary lifestyle, defined as engaging in less than 60 minutes of regular physical training per week during the previous six months
* No prior experience in wrestling or any other organized combat sports
* Healthy with no known medical conditions that could interfere with participation

Exclusion Criteria:

* Respiratory disease (chronic or acute)
* Musculoskeletal injuries that could impede training participation
* Chronic illnesses requiring ongoing medical treatment
* Diagnosed psychological disorders that could affect their ability to safely engage in physical activity

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
WHO-5 Well-Being Index | 6 week
  The WHO-5 Well-Being Index is a brief global measure of current psychological well-being. It consists of five positively phrased items that reflect mood, vitality, and general life satisfaction.
Sport Anxiety Scale-2 (SAS-2) | 6 week
  The Sport Anxiety Scale-2 (SAS-2) was used to assess multidimensional components of sport-related anxiety. The scale includes 15 items scored on a 4-point Likert scale (1 = not at all, 4 = very much).

SECONDARY OUTCOMES:
Brief Psychological Resilience Scale (BPRS) | 6 week
  The Brief Psychological Resilience Scale (BPRS) evaluates an individual's capacity to "bounce back" or recover quickly from stressful situations. It includes 6 items rated on a 5-point Likert scaleintervention
Body composition measurement | 6 weeks
  In the study, body composition (e.g., body fat percentage and muscle mass) was assessed using a Jawon Medical GAIA 359 Plus bioelectrical impedance analyzer (Jawon Medical Co., South Korea), with data managed through the BodyPass software (GAIA 359 Plus version). This device was used to confirm that all participants had comparable baseline body characteristics. Body weight was recorded using the same analyzer, while height (cm) was measured with a portable stadiometer

CONTACTS AND LOCATIONS:
Overall Officials: coşkun yılmaz, associate professor, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF